CLINICAL TRIAL: NCT04734210
Title: A Multicenter, Randomized, Double-Masked, Dose-Ranging Study To Compare The Ocular Safety, Tolerability, And Efficacy Of SURF-200 Ophthalmic Solution (0.02% And 0.04% Betamethasone Sodium Phosphate) To Vehicle In Subjects With A Diagnosis Of Dry Eye Disease And Experiencing An Episodic Flare Up
Brief Title: Research Study To See How Well An Eye Drop (SURF-200) Works, What Side Effects There Are, And To Compare It With Vehicle In Subjects With An Episodic Flare-Up of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Surface Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-200-001
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — betamethasone sodium phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SURF-200 (0.02% betamethasone sodium phosphate in vehicle) (Experimental): One drop twice daily (BID) in the study eye for 14 days.
  Interventions: Drug: 0.02% Betamethasone Sodium Phosphate
- SURF-200 (0.04% betamethasone sodium phosphate in vehicle) (Experimental): One drop BID in the study eye for 14 days.
  Interventions: Drug: 0.04% Betamethasone Sodium Phosphate
- Vehicle (Placebo Comparator): One drop BID in the study eye for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.02% Betamethasone Sodium Phosphate — topical corticosteroid solution
  Arms: SURF-200 (0.02% betamethasone sodium phosphate in vehicle)
Drug: 0.04% Betamethasone Sodium Phosphate — topical corticosteroid solution
  Arms: SURF-200 (0.04% betamethasone sodium phosphate in vehicle)
Drug: Placebo — topical vehicle solution
  Arms: Vehicle

SUMMARY:
SURF-200 is being studied in people experiencing an episodic flare-up of their dry eye disease. SURF-200 is an investigational drug (which means the study drug is currently being tested) in the form of a sterile eye drop.

The purpose of this research study is to see how well SURF-200 works and what side effects there are, and to compare it with vehicle (placebo). The study will involve about 120 study participants at multiple research sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older who have a diagnosis of dry eye disease and experiencing an episodic flare up. Criteria for the diagnosis must include the following:

   1. UNC DEMS score of greater than or equal to 5 but less than or equal to 9
   2. Conjunctival hyperemia score of greater than or equal to 2 in the study eye when using the conjunctival hyperemia reference photos
   3. Schirmer's Tear Test score (with anesthesia) greater than 1 mm but less than or equal to12 mm in the study eye
2. Subjects must be able to understand and sign the Informed Consent Form (ICF).
3. Female subjects of childbearing potential must agree to and submit a negative urine pregnancy test before any study-specific procedures are performed. The subjects must be using and continue to use a suitable method of contraception for the duration of the study: spermicide with barrier, oral contraceptive, transdermal contraceptive, injectable or implantable contraceptive, intrauterine device (IUD), abstinence or surgical sterilization of a partner. If a subject is not of childbearing potential (e.g., has been postmenopausal for at least 12 months or is premenarchal, or has undergone a hysterectomy, bilateral oophorectomy or a bilateral tubal ligation), a urine pregnancy test and use of a suitable method of contraception for the duration of the study will not be required.
4. Subjects must have a best-corrected visual acuity (BCVA) of at least +1.0 log of the minimum angle of resolution (logMAR) (Snellen equivalent of 20/200) in the non-study eye (fellow eye).
5. Subjects must have an intraocular pressure (IOP) of >8 mmHg and ≤22 mmHg in the study eye.
6. Subjects who are on Restasis, Xiidra or other cyclosporine ophthalmic eye drops must be on a stable dose for at least 4 months prior to Screening Visit 1 (Day -14 to Day 0) and remain compliant with the use of these medications throughout the duration of this study.
7. Subjects who are on artificial tears, oral antihistamines, beta blockers and diuretics must be on a stable dose for at least 1 month prior to Screening Visit 1 (Day -14 to Day 0) and remain compliant with the use of these medications throughout the duration of this study.
8. Subjects must be willing and able to attend all study visits and follow all instructions.
9. Subjects must be able to self-instill the study drug (if unable, a caregiver must be available to instill all doses of the study drug).
10. Have a history of use or desire to use an eye drop for dry eye symptoms for longer than the past 6 months.

Exclusion Criteria:

1. Females who are pregnant or nursing or planning to become pregnant during the study. Females of childbearing potential (not surgically sterilized or postmenopausal) may not participate in the study if they do not agree to use adequate birth control methods for the duration of the study.
2. Use of contact lenses in either eye during the study. Contact lens wear must have been discontinued at least 2 weeks prior to Baseline/Randomization Visit 2 (Day 1).
3. Use of corticosteroids or nonsteroidal anti-inflammatory agents (NSAID) (except oral doses of aspirin at 81 mg/day or lower) within 2 weeks of the initiation of study drug at Baseline/Randomization Visit 2 (Day 1) and for the remainder of the study.
4. Inhaled, ingested, sublingual, transdermal or topical products containing marijuana, tetrahydrocannabinol (THC) or cannabidiol (CBD) within 7 days of the first dose of study drug at Baseline/Randomization Visit 2 (Day 1) and for the remainder of the study.
5. Presence or history of treatment with systemic immunosuppressive or chemotherapeutic agents.
6. History of high IOP response to steroids.
7. Participated in an ophthalmic investigational product clinical trial within 30 days of Screening Visit 1 (Day -14 to Day 0).
8. Active collagen vascular disorder or autoimmune disease.
9. A condition or a situation, which in the investigator's opinion may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.
10. Known hypersensitivity to any component of the study drug or procedural medications.
11. Known hypersensitivity to steroids.
12. Any active corneal epithelial/stromal pathology noted in the study eye at Screening Visit 1 (Day -14 to Day 0).
13. Any history of corneal surgery in the study eye (including corneal crosslinking, radial keratotomy, corneal transplant, or LASIK).
14. Any ocular surgery in the study eye within the past year.
15. Subject has punctal occlusion with any modality or a change in punctal plug status in either eye within the 3 months prior to Screening Visit 1 (Day -14 to Day 0).
16. Subject has a history of glaucoma.
17. Subject has a history of herpes simplex infection in either eye.
18. Subject has active corneal, conjunctival or canalicular pathology (including ocular infection [bacterial, viral or fungal]) in either eye. Specifically, active viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, and mycobacterial infection of either eye and fungal diseases of the ocular structures (such as fungal keratitis).
19. Subject has thinning of the cornea or sclera in the study eye.
20. Subject has active anterior blepharitis in the study eye.
21. Subject has a history of uveitis in the study eye.
22. Subject is suffering from alcohol and/or drug abuse.
23. Subject has tested positive for the COVID-19 virus within 30 days prior to Screening Visit 1 (Day -14 to Day 0).
24. Subject has previously received treatment in this study protocol.
25. Subject is taking a medication, that in the opinion of the investigator, might interfere with the study parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Hosseini, MD, PhD, Study Chair — Surface Ophthalmics, Inc. (formerly Surface Pharmaceuticals, Inc.)
Locations (28):
- United States (28):
  - Trinity Research Group, Dothan, Alabama
  - Canyon City EyeCare, Azusa, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Visionary Eye Institute, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Vision Institute, Colorado Springs, Colorado
  - The Eye Center of Northern Colorado, Fort Collins, Colorado
  - Connecticut Eye Consultants, PC, Danbury, Connecticut
  - The Eye Associates of Manatee, Bradenton, Florida
  - Blue Ocean Clinical Research (The Macula Center), Clearwater, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Eye Center of North Florida PA, Panama City, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Chu Vision Institute, Bloomington, Minnesota
  - Complete Eye Care, Hamel, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Consultants Ltd., St Louis, Missouri
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Total Eye Care, PA, Memphis, Tennessee
  - West TN EyeCare dba Toyos Clinic, Nashville, Tennessee
  - Advanced Laser Vision & Surgical Institute, Houston, Texas
  - R and R Eye Research, LLC, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study periods:
  Dosing Days 1-14.
  Follow-up (FU) to Day 28: Responders continued in the study; non-responders discontinued. Responders had to have a reduction of ≥1 unit in UNC DEMS score and a ≥0.5 point reduction in conjunctival hyperemia grade (study eye) compared to baseline.
  FU to Day 70 or rebound: Responders were followed up to Day 70 or rebound. Rebound was defined as worsening in UNC DEMS score of ≥1 unit and a worsening in conjunctival hyperemia of ≥0.5 point (study eye).
Pre-assignment Details: Prior to each participant's assignment by chance to one of the three treatment arms/groups (randomization), the Investigator designated the participant's Study Eye. The participant's Study Eye was the eye that was eligible for the study and had the worst signs and symptoms. The participant's other eye was called the Fellow Eye.
Units Other Than Participants: Study eyes
Groups:
- SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle): Eye Drops: 0.02% Betamethasone Sodium Phosphate (topical corticosteroid solution)
  Dosing: One drop twice daily in the study eye for 14 days.
- SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle): Eye drops: 0.04% Betamethasone Sodium Phosphate (topical corticosteroid solution)
  Dosing: One drop twice daily in the study eye for 14 days.
- Vehicle: Eye drops: Placebo (topical vehicle solution)
  Dosing: One drop twice daily in the study eye for 14 days.
Period: Two-week Dosing Period (Days 1 - 14)
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Started | 47; 47 Study eyes | 45; 45 Study eyes | 47; 47 Study eyes
Completed | 44; 44 Study eyes | 44; 44 Study eyes | 46; 46 Study eyes
Not Completed | 3; 3 Study eyes | 1; 1 Study eyes | 1; 1 Study eyes
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Did not complete dosing with study drug but remained in the study for safety follow-up at Day 28. | 1 | 0 | 0
Not completed — Did not dose with study drug; missed Day 8 visit and did not return dosing diary. Lost to follow-up. | 0 | 0 | 1
Period: Safety Follow-up to Day 28
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Started | 44; 44 Study eyes | 44; 44 Study eyes | 46; 46 Study eyes
Completed | 30; 30 Study eyes | 34; 34 Study eyes | 30; 30 Study eyes
Not Completed | 14; 14 Study eyes | 10; 10 Study eyes | 16; 16 Study eyes
Period: Safety Follow-up to Day 70 or Rebound
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Started | 30; 30 Study eyes | 34; 34 Study eyes | 30; 30 Study eyes
Completed | 24; 24 Study eyes | 24; 24 Study eyes | 25; 25 Study eyes
Not Completed | 6; 6 Study eyes | 10; 10 Study eyes | 5; 5 Study eyes

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: It included all randomized subjects regardless of whether post-baseline measures were collected, or study drug was received.
Units Other Than Participants: Study Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle | Total
Number analyzed (Participants) | 47 | 45 | 47 | 139
Number analyzed (Study Eyes) | 47 | 45 | 47 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (15.9) | 60.9 (14.1) | 59.7 (15.3) | 60.2 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 37 | 106
  Male | 12 | 11 | 10 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 13 | 41
  Not Hispanic or Latino | 33 | 30 | 32 | 95
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 4 | 14
  White | 41 | 40 | 39 | 120
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
University of North Carolina Dry Eye Management Scale (UNC DEMS) Score at Baseline [Mean (Standard Deviation); unit: UNC DEMS units] — The UNC DEMS scale is a participant-specific 10-point scale with a minimum score of 1 ([1-2] My symptoms are not a problem. My dry eye does not affect my daily life at all) and a maximum score of 10 ([9-10] my symptoms are severe and I need immediate medical care. My dry eye greatly affects my daily life).
  UNC DEMS units | 6.9 (1.2) | 7.2 (1.1) | 6.9 (1.2) | 7.0 (1.1)
Conjunctival hyperemia score in study eye at baseline [Mean (Standard Deviation); unit: units on a scale] — Conjunctival hyperemia was graded by Investigator using the scale below and clinical grade reference photos:
  Grade 0 (none: no hyperemia of the bulbar conjunctiva)
  Grade 0.5 (Grade 0 plus dilation of at least a couple of conjunctival blood vessels [CBVs] but less than Grade 1)
  Grade 1 (mild: the dilation of a few CBVs)
  Grade 1.5 (Grade 1 plus dilation of some CBVs but less than Grade 2)
  Grade 2 (moderate: the dilation of several CBVs)
  Grade 2.5 (Grade 2 plus dilation of many CBVs but less than Grade 3)
  Grade 3 (severe: the abundant and overwhelming dilation of many CBVs)
  units on a scale | 2.2 (0.4) | 2.3 (0.4) | 2.4 (0.4) | 2.3 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: University of North Carolina Dry Eye Management Scale (UNC DEMS) Responder Analysis
Description: The UNC DEMS scale is a participant-specific 10-point scale with a minimum score of 1 ([1-2] My symptoms are not a problem. My dry eye does not affect my daily life at all) and a maximum score of 10 ([9-10] my symptoms are severe and I need immediate medical care. My dry eye greatly affects my daily life).
  Participants with a minimum reduction of ≥1 point in UNC DEMS score from baseline were defined as responders, and response rates were summarized by treatment group.
Time Frame: Baseline and Day 8
Population: Intent-to-Treat (ITT) Population: included all randomized subjects regardless of whether post-baseline measures were collected, or study drug was received. For the ITT responder analysis, the analysis was conducted based on the observed available data without any imputation for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Number analyzed (Participants) | 47 | 45 | 46
percentage of responders | 53.2 [38.1 to 67.9] | 60.0 [44.3 to 74.3] | 65.2 [49.8 to 78.6]
Statistical Analysis 1: Comparison: SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) vs SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) vs Vehicle; Exploratory Phase 2 Study; approximately 120 subjects (approximately 40 subjects per each of the 3 treatment groups) were planned to be enrolled in the study. The sample size was based on medical judgment. No formal sample size calculation was performed, and the sample size was empirical. However, the sample size selected was considered sufficient to adequately characterize the general safety and efficacy profile of the study treatments; Test type: Other — Exploratory, descriptive analysis; p = 0.2933, Fisher Exact — The difference in response rates between each of the SURF-200 formulations and vehicle was compared by Fisher's exact method; The threshold for statistical significance is p=0.05

2. Secondary Outcome: University of North Carolina Dry Eye Management Scale (UNC DEMS) Responder Analysis
Description: as for outcome 1
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Number analyzed (Participants) | 45 | 44 | 45
percentage of responders | 88.9 [75.9 to 96.3] | 93.2 [81.3 to 98.6] | 82.2 [67.9 to 92.0]
Statistical Analysis 1: Comparison: SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) vs SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) vs Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Exploratory, descriptive analysis; p = 0.1966, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; The threshold for statistical significance is p=0.05

3. Secondary Outcome: Conjunctival Hyperemia Responder Analysis
Description: Conjunctival hyperemia was graded by Investigator using the scale below and clinical grade reference photos:
  Grade 0 (none: no hyperemia of the bulbar conjunctiva)
  Grade 0.5 (Grade 0 plus dilation of at least a couple of conjunctival blood vessels [CBVs] but less than Grade 1)
  Grade 1 (mild: the dilation of a few CBVs)
  Grade 1.5 (Grade 1 plus dilation of some CBVs but less than Grade 2)
  Grade 2 (moderate: the dilation of several CBVs)
  Grade 2.5 (Grade 2 plus dilation of many CBVs but less than Grade 3)
  Grade 3 (severe: the abundant and overwhelming dilation of many CBVs)
  Participants with a minimum reduction of ≥0.5 point in conjunctival hyperemia grade in the study eye from baseline were defined as responders, and response rates were summarized by treatment group.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle): Eye drops: 0.04% Betamethasone Sodium Phosphate (topical corticosteroid solution)
  Dosing: One drop BID in the study eye for 14 days.
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
Number analyzed (Participants) | 47 | 45 | 46
percentage of responders | 38.3 [24.5 to 53.6] | 62.2 [46.5 to 76.2] | 37.0 [23.2 to 52.5]
Statistical Analysis 1: Comparison: SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) vs SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) vs Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Exploratory, descriptive analysis; p = 0.0213, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; The threshold for statistical significance is p=0.05

ADVERSE EVENTS:
Time Frame: From each participant's signature of informed consent at Screening through Day 70 (completion of the study) or early withdrawal, which ever came first.
Description: Adverse events were collected systematically at each study visit, from each participant's signature of informed consent at Screening through Day 70 (completion of the study) or early withdrawal.
Arm/Group | SURF-200 (0.02% Betamethasone Sodium Phosphate in Vehicle) | SURF-200 (0.04% Betamethasone Sodium Phosphate in Vehicle) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 0/47 | 0/45 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04734210/Prot_SAP_000.pdf